CLINICAL TRIAL: NCT00367029
Title: Achieving Physical Activity Guidelines Through an Enhanced Print Intervention
Brief Title: Individualized Motivational Print Materials to Encourage More Physical Activity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: The Miriam Hospital, Centers for Behavioral and Preventive Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 408; R01HL064342-05 (NIH)
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Print-based, individually tailored motivational program
  Interventions: Behavioral: Individualized Print-Based Motivational Program
- 2 (Experimental): Enhanced version of the print-based, individually tailored motivational program
  Interventions: Behavioral: Individualized Print-Based Motivational Program

INTERVENTIONS:
Behavioral: Individualized Print-Based Motivational Program — Study researchers will develop individualized reports, manuals, and tip sheets that include feedback and strategies for increasing physical activity for each participant. Materials will be mailed to participants 14 times throughout the year.
  Participants in the enhanced intervention will receive additional materials that focus on increasing social support, self regulation, and outcome expectations, as well as materials on how to effectively monitor physical activity levels. They will also attend one study visit to assess their goals with the research staff.

SUMMARY:
Individuals who are not physically active are at risk for developing heart disease, stroke, and diabetes. Using motivational print materials is one way to encourage individuals to increase their physical activity. This study will evaluate the effect that an enhanced version of an individualized, print-based motivational program has on increasing physical activity among sedentary individuals.

DETAILED DESCRIPTION:
Currently, only 32% of adults in the United States participate in regular physical activity. Several healthcare organizations, including the Centers for Disease Control and Prevention, the National Institutes of Health, and the American Heart Association recommend that adults engage in a minimum of 2 ½ hours of physical activity each week. In a previous study, individuals who received motivational print materials in the mail increased their weekly physical activity more than individuals who received no motivational materials or who received motivational support over the telephone. However, about half of those who were mailed the print materials still did not reach the recommended goal of 2 ½ hours of physical activity per week. The purpose of this study is to compare the effectiveness of an enhanced version of an individualized, print-based motivational program versus a previously tested print-based motivational program at increasing physical activity levels in sedentary individuals.

This study will enroll healthy, sedentary individuals. Participants will be randomly assigned to either a print-based, individually tailored motivational program or an enhanced version of the same program. All participants will attend a baseline study visit, which will include body measurements, physical activity assessments, and health and psychological questionnaires. A select group of participants will also take part in an exercise test. Participants will then document their monthly physical activity. Study researchers will use this information, as well as the completed questionnaires, to develop individualized reports, manuals, and tip sheets that include feedback and strategies for increasing physical activity for each participant. Materials will be mailed to participants 14 times throughout the year. Participants in the enhanced intervention will receive additional materials that focus on increasing social support, self regulation, and outcome expectations, as well as materials on how to effectively monitor physical activity levels. They will also attend one study visit to assess their goals with the research staff. At Months 6 and 12, baseline evaluations will be repeated and all participants will be interviewed to assess physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Sedentary
* Able to speak and read English
* Planning to live in the area for the duration of the study

Exclusion Criteria:

* Currently participates in 91 or more minutes of moderate or vigorous physical activity per week
* Heart disease
* Cerebrovascular disease
* Peripheral vascular disease
* Chronic obstructive pulmonary disease
* Diabetes
* High blood pressure
* History of gastric bypass surgery
* Psychoses
* Any serious medical problem that would make exercise unsafe or unwise
* Prior participation in a hospital-based or medically supervised weight loss program
* Excessive alcohol consumption
* Pregnant or plans to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2006-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Achievement of 150 minutes per week of at least moderate intensity physical activity | Measured by the 7-day Physical Activity Recall test at Months 6 and 12

SECONDARY OUTCOMES:
Moderators and mediators of the intervention (e.g., motivation and enjoyment) | Measured at Months 6 and 12
Cost-effectiveness | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Bess H. Marcus, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Centers for Behavioral and Preventive Medicine, The Miriam Hospital, Providence, Rhode Island, United States